CLINICAL TRIAL: NCT02444338
Title: Randomised Investigation of the MitraClip Device in Heart Failure: 2nd Trial in Patients With Clinically Significant Functional Mitral Regurgitation
Brief Title: A Clinical Evaluation of the Safety and Effectiveness of the MitraClip System in the Treatment of Clinically Significant Functional Mitral Regurgitation
Acronym: Reshape-HF2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Goettingen (Other)
Responsible Party: Principal Investigator, Karsten Gavenis, on behalf of Principle Investigator Prof. Wolfgang Schillinger and Prof. Stefan D. Anker, University Medical Center Goettingen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Version No. 6.0
Record Dates: First submitted 2015-05-12; First posted 2015-05-14 (Estimated); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Mitral Valve Insufficiency
MeSH Terms: conditions — Mitral Valve Insufficiency | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: PROBE
  * outcome assessment: blinded
  * patient & investigator: open
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Group (Active Comparator): optimal standard of care therapy
  Interventions: Other: standard of care
- Device Group (Experimental): MitraClip device plus optimal standard of care therapy
  Interventions: Device: MitraClip; Other: standard of care

INTERVENTIONS:
Device: MitraClip — Implantation of the MitraClip System for patients with chronic heart failure.
  Arms: Device Group
Other: standard of care

SUMMARY:
To study the safety and effectiveness of the MitraClip System in the treatment of clinically significant functional mitral regurgitation in patients with New York Heart Association (NYHA) Functional Class II to Class IV chronic heart failure.

DETAILED DESCRIPTION:
The trial is designed to provide additional evidence regarding appropriate recommendations for use of the MitraClip System for patients with chronic heart failure and clinically significant functional mitral regurgitation. Additionally, the trial will collect evidence regarding health economics of the MitraClip System for use in this patient population.

ELIGIBILITY:
Key Inclusion Criteria:

* Clinically significant functional mitral regurgitation (moderate-to-severe or severe MR) as defined by European Association of Echocardiography, within 90 days prior to randomization and confirmed by the Echocardiography Core Laboratory Note: The TTE must be obtained after the subject has been stabilized on optimal therapy and has undergone revascularization and/or CRT, as appropriate
* Assessed by the investigator to be on optimal standard of care therapy for heart failure, according to current ESC/HFA guidelines with no dose changes of heart failure drugs (with the exception of diuretics) during the last 2 weeks immediately prior to randomization.
* Symptomatic with documented New York Heart Association Class II, III or IV heart failure, despite optimal standard of care therapy, within 30 days preceding randomization
* Minimum of one documented hospitalization (acute care admission or emergency room visit) for heart failure within 12 months preceding randomization OR values of 300 pg/mL for BNP or 1000 pg/mL for NT-proBNP after optimal medical and/or device management within 90 days preceding randomization Note: BNP or NT-proBNP must be obtained after the subject has been stabilized on optimal therapy and has undergone revascularization and/or CRT, as appropriate
* Ambulatory patient with symptomatic congestive heart failure (CHF) in NYHA functional class II to IV (despite optimal standard of care therapy as assessed within 30 days preceding randomization) and with LVEF 20% to 50%. Note: LVEF needs to be determined by one of the following methods: transthoracic echocardiography (TTE), contrast ventriculography, gated blood pool scan, cardiac magnetic resonance) within 90 days prior to randomization
* Patient is ambulatory and able to perform a 6MWT with the only limiting factor(s) being due to cardiovascular fitness

Key Exclusion Criteria:

* Mitral regurgitation is primarily due to degenerative disease of the mitral valve apparatus (Degenerative MR) as determined by transesophageal echocardiography (TEE).
* Status 1 heart transplant or prior orthotropic heart transplantation.
* Introduction of a new heart failure drug class within the last 2 weeks prior to randomization.
* Evidence of acute coronary syndrome, transient ischemic attack or stroke within 90 days prior to randomization. Note:Acute coronary syndrome (ACS) is defined as an ACS that requires an intervention. Increased troponin without acute symptoms and chest pain is not defined as ACS.
* Any percutaneous cardiovascular intervention, carotid surgery, cardiovascular surgery, or atrial fibrillation ablation within 90 days prior to randomization.
* Therapy with or without cardioverter-defibrillator (CRT or CRT-D), or Implantable Cardioverter Defibrillator (ICD)) within 90 day prior to randomization, or revision of any implanted rhythm management device within 90 days prior to randomization.
* Need for any cardiovascular surgery.
* Mitral valve surgery is considered the preferred therapeutic option for the subject
* Renal replacement therapy
* 6-Minute Walk Test (6MWT) distance > 475 meters
* Mitral Valve Area (MVA) by planimetry < 4.0 cm2; if MVA by planimetry is not measurable, pressure half-time measurement is acceptable; MVA must be confirmed by the Echocardiography Core Laboratory

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 505 (Actual)
Dates: Start 2015-03; Primary Completion 2024-04-19 (Actual); Study Completion 2024-04-19 (Actual)

PRIMARY OUTCOMES:
Composite rate of recurrent heart failure hospitalizations and cardiovascular (CV) death within 24 months | 24 months
  Composite rate of recurrent heart failure hospitalizations and cardiovascular (CV) death within 24 months
Rate of total (first and recurrent) HF hospitalizations within 24 months | 24 months
  Rate of total (first and recurrent) HF hospitalizations within 24 months
Change in quality of life (i.e. overall KCCQ score) from baseline to 12 months | 12 months
  Change in quality of life (i.e. overall KCCQ score) from baseline to 12 months

SECONDARY OUTCOMES:
Percentage of patients with mitral regurgitation grade of 2+ or lower at 12 months as assessed by the Echocardiography Core Laboratory | at 12 months
  Percentage of patients with mitral regurgitation grade of 2+ or lower at 12 months as assessed by the Echocardiography Core Laboratory
Change in 6 Minute Walking Test distance from baseline to 12 months | from baseline to 12 months
  Change in 6 Minute Walking Test distance from baseline to 12 months
All-cause mortality during all available follow-up | during all available follow-up
  All-cause mortality during all available follow-up
Rate of total (first and recurrent) hospitalizations for any cause within 24 months | 24 months
  Rate of total (first and recurrent) hospitalizations for any cause within 24 months
Percentage of patients in NYHA function class I/II at 12 months | 12 months
  Percentage of patients in NYHA function class I/II at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Schillinger, Prof., Principal Investigator — University Medical Center Göttingen
Locations (35):
- Klinika Kardiologie IKEM, Prague, Czechia
- Denmark (2):
  - Rigshospitalet Copenhagen, Copenhagen
  - OUH Odense, Odense
- Germany (10):
  - Charité, Berlin
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Universitätsklinikum Essen, Essen
  - Johanniter Krankenhaus, Genthin
  - University Medical Center Goettingen, Göttingen
  - Universitätsklinikum Halle, Halle
  - University Hospital Heidelberg, Heidelberg
  - Universitätsklinikum Jena, Jena
  - University Hospital Mainz, Mainz
  - Universitätsklinik Würzburg, Würzburg
- Greece (3):
  - HYGEIA Hospital Athens, Athens
  - Interbalkan Medical Center, Thessaloniki
  - St. Luke's Hospital Thessaloniki, Thessaloniki
- AOC Brescia, Brescia, Italy
- Poland (5):
  - Cardiology Department at Samodzielny Publiczny Szpital Kliniczny nr 7, Katowice
  - Krakowski Szpital Specjalistyczny im. Jana Pawła II, Krakow
  - Poznan Medical University, Poznan
  - Medical University Department of Heart Diseases, Wroclaw
  - Śląskie Centrum Chorób Serca, Zabrze
- Portugal (3):
  - Lisbon St. Marta Hospital, Lisbon
  - Lisbon St. Maria Hospital, Lisbon
  - Centro Hospitalar Vila Nova de Gaia / Espinho, Vila Nova de Gaia
- Spain (4):
  - Hospital Germans Trias i Pujol, Badalona
  - HUL Leon, León
  - Hospital Universitario Central de Asturias, Oviedo
  - Instituto de Ciencias del Corazón (ICICOR), Valladolid
- United Kingdom (6):
  - Royal Infirmary of Edinburgh, Edinburgh
  - Golden Jubilee National Hospital, Glasgow
  - Castle Hill Hospital, Hull
  - The Royal Brompton and Harefield Hospitals, London
  - Wythenshawe Hospital of South Manchester - Manchester University NHS Foundation Trust (MFT), Manchester
  - Royal Stoke Hospital - University Hospital of North Midlands, Stoke-on-Trent

REFERENCES:
- [Result] Anker SD, Friede T, von Bardeleben RS, Butler J, Khan MS, Diek M, Heinrich J, Geyer M, Placzek M, Ferrari R, Abraham WT, Alfieri O, Auricchio A, Bayes-Genis A, Cleland JGF, Filippatos G, Gustafsson F, Haverkamp W, Kelm M, Kuck KH, Landmesser U, Maggioni AP, Metra M, Ninios V, Petrie MC, Rassaf T, Ruschitzka F, Schafer U, Schulze PC, Spargias K, Vahanian A, Zamorano JL, Zeiher A, Karakas M, Koehler F, Lainscak M, Oner A, Mezilis N, Theofilogiannakos EK, Ninios I, Chrissoheris M, Kourkoveli P, Papadopoulos K, Smolka G, Wojakowski W, Reczuch K, Pinto FJ, Wiewiorka L, Kalarus Z, Adamo M, Santiago-Vacas E, Ruf TF, Gross M, Tongers J, Hasenfuss G, Schillinger W, Ponikowski P; RESHAPE-HF2 Investigators. Transcatheter Valve Repair in Heart Failure with Moderate to Severe Mitral Regurgitation. N Engl J Med. 2024 Nov 14;391(19):1799-1809. doi: 10.1056/NEJMoa2314328. Epub 2024 Aug 31. PMID 39216092
- [Result] Anker SD, Friede T, von Bardeleben RS, Butler J, Fatima K, Diek M, Heinrich J, Hasenfuss G, Schillinger W, Ponikowski P. Randomized investigation of the MitraClip device in heart failure: Design and rationale of the RESHAPE-HF2 trial design. Eur J Heart Fail. 2024 Apr;26(4):984-993. doi: 10.1002/ejhf.3247. Epub 2024 Apr 23. PMID 38654139
- [Derived] McMurray JJV, Metra M. Transcatheter Repair of Secondary Mitral Regurgitation. N Engl J Med. 2023 Jun 1;388(22):2097-2098. doi: 10.1056/NEJMe2302924. No abstract available. PMID 37256981